CLINICAL TRIAL: NCT03567980
Title: A Proof of Concept Clinical Trial Evaluating the Safety and Efficacy of Eucrisa (Crisaborole) in Patients With Seborrheic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Boni Elewski, Professor and Chair, UAB Department of Dermatology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180306
Record Dates: First submitted 2018-06-11; First posted 2018-06-26 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — crisaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- topical crisaborole 2% (Experimental)
  Interventions: Drug: Crisaborole

INTERVENTIONS:
Drug: Crisaborole — Application of topical crisaborole 2% ointment on the face for 4 weeks to evaluate the anti-inflammatory action of this agent and its utility in the treatment of facial seborrheic dermatitis.

SUMMARY:
Seborrheic dermatitis is a common and recurrent dermatosis that characteristically involves the scalp, nasolabial folds, eyebrows, glabella, and upper eye lids. It presents as an erythematous, thin scaly patch with a greasy sandpaper texture that varies depending on disease severity. While seborrheic dermatitis most frequently occurs on the face, it can involve other areas of the body especially the chest, abdomen, and axilla. Overall incidence is thought to be between 2-5% of the general population, though this is likely an underestimation. Pruritus is variable, though the signs and symptoms of this disorder are certainly worsened by certain external conditions especially weather, personal perspiration, stress, and poor hygiene. Patients often complain about the red, scaly patches on the face.

Antifungal agents are frequently used as monotherapy or in combination regimens in the treatment of seborrheic dermatitis. Topical corticosteroids are often used for their anti-inflammatory effects. Long term use of topical steroids on the face is not a preferred treatment modality due to the risk of striae development and other textural changes that occur over time. Therefore, topical crisaborole may be an alternative given its non-corticosteroid anti-inflammatory action. Crisaborole is a phosphodiesterase-4 (PDE-4) inhibitor that increases intracellular cyclic AMP (cAMP) levels to exert its anti-inflammatory effects. While it has not previously been investigated for its effects in seborrheic dermatitis, further studies evaluating its role in this disease are warranted.

Therefore, the investigators propose a proof of concept study using topical crisaborole 2% ointment on the face for 4 weeks to evaluate the anti-inflammatory action of this agent and its utility in the treatment of facial seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed.
2. Male or female subjects 18 to 70 years of age.
3. Able to complete the study and to comply with study instructions.
4. Female subjects of childbearing potential must have a negative pregnancy test. Sexually active women of childbearing potential participating in the study must agree to use a medically acceptable form of contraception (which includes oral contraception, injectable or implantable methods, or intrauterine devices) during the entire duration of the study
5. Mild to moderate seborrheic dermatitis on the face with an ISGA of 2 or 3 at baseline.

Exclusion Criteria:

1. Use of systemic antifungal agents, corticosteroids or other immunosuppressive therapies, or systemic retinoids within 4 weeks prior to the baseline visit.
2. Use of topical antifungal therapy, corticosteroid therapy, or calcineurin inhibitors to the face, within 2 weeks prior to the baseline visit. Topical, over-the-counter antifungal shampoo will be allowed as long as it has remained constant for 4 weeks prior to baseline.
3. Use of any investigational drugs within 4 weeks prior to the baseline visit, or subjects scheduled to receive an investigative drug other than the study product during the period of the study.
4. History of known or suspected intolerance to any of the ingredients of the study product.
5. Female subjects who are pregnant, trying to become pregnant or lactating.
6. Any clinically relevant abnormal vital signs or findings on the physical examination which in the opinion of the investigator might interfere with the study assessments.
7. A clinically relevant history of abuse of alcohol or other drugs.
8. Any major illness within 30 days prior to the baseline visit.
9. Subjects with any clinically significant condition which would, in the opinion of the investigator, compromise the subject's participation in the study.
10. Subjects who are immunocompromised (ex: HIV).
11. Considered unable or unlikely to attend the necessary visits.
12. Currently using any medication, which in the opinion of the investigator may affect the evaluation of the study product
13. Subjects who have significant neurological conditions (Parkinson's disease or Stroke), who in the opinion of the investigator are not eligible for the study due to the severity of neurological condition.
14. Subjects with a history of non-melanoma skin cancer of the face within 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Dermatology at the Whitaker Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical Crisaborole 2%
Started | 30
Completed | 29
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Topical Crisaborole 2%
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (3.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 16
  White | 14
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in ISGA (Investigator's Static Global Assessment) Score
Description: • Investigator's Static Global Assessment (ISGA) is a skin assessment tool utilized in clinical trials. The tool is based on a 5-point scale with 0 or 1 (clear or almost clear) being the best score one could receive, while a score of 4 is the worst score available and indicates severe disease. ISGA will be collected via skin examination to evaluate efficacy of Crisaborole 2% topical ointment in the treatment of seborrheic dermatitis. A 0 or 1 (clear or almost clear) on the ISGA would be considered a treatment success. Percent change in ISGA score from baseline to 4 weeks will be measured and reported.
Time Frame: Baseline to 4 weeks
Population: One participant withdrew due to adverse events (headaches and facial pain)
Measure: Number; unit: percent change
Arm/Group | Topical Crisaborole 2%
Number analyzed (Participants) | 29
percent change | 67.8

2. Secondary Outcome: Itch NRS (Itch Numeric Rating Scale)
Description: • The Itch Numeric Rating Scale (NRS) is a subject-administered, 11 point horizontal scale anchored at 0 and 10, 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a subject itching is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
  The Itch NRS (A numeric measurement of itch) will be collected to assess the percentage of improvement of patient reported itching. This will be calculated as a percent changes from baseline in the Itch NRS scale.
Time Frame: Baseline to 4 weeks
Population: One participant withdrew due to adverse events (headaches and facial pain)
Measure: Number; unit: percent change
Arm/Group | Topical Crisaborole 2%
Number analyzed (Participants) | 29
percent change | 45

3. Other Pre Specified Outcome: Number of Participants With Adverse Events That Are Related to Treatment.
Time Frame: Baseline to 4 weeks
Population: All enrolled patients were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Crisaborole 2%
Number analyzed (Participants) | 30
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the screening visit to the end of study visit for each participant, a total of 4 weeks per participant evaluation.
Arm/Group | Topical Crisaborole 2%
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Crisaborole 2% (N=30)
Headaches (General disorders) | 1 (1)
Facial Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03567980/Prot_SAP_000.pdf